CLINICAL TRIAL: NCT03979183
Title: 'Physio-EndEA' Study: a Randomized Controlled Trial to Evaluate the Effect of a Supervised and Adapted Rehabilitation Program to Improve Quality of Life in Women Diagnosed With Endometriosis
Brief Title: Effect of a Rehabilitation Program to Improve Quality of Life in Women Diagnosed With Endometriosis (Physio-EndEA Study)
Acronym: Physio-EndEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Artacho Cordón, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Physio-EndEA
Record Dates: First submitted 2018-07-10; First posted 2019-06-07 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Endometriosis
Keywords: Pain; Therapeutic exercise; Physiotherapy; Rehabilitation; Quality of life
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Therapeutic exercise
  Interventions: Behavioral: Lumbopelvic, stretching, aerobic and relaxation exercises
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Lumbopelvic, stretching, aerobic and relaxation exercises — Intervention program will comprises brisk walks and small choreographies, global and analytical stretching exercises, as well as lumbopelvic stabilization exercises (with intensity and volume progression)
  Arms: Intervention

SUMMARY:
Given (1) the high volume of women on reproductive age that have a clinical diagnosis of endometriosis and (2) the poor management of symptoms that medical treatment usually achieves, new therapeutic interventions need to be evaluated in order to improve pain and quality of life in those patients. Therefore, 'Physio-EndEA' study has been designed to evaluate whether therapeutic exercise could help on the management of endometriosis-related symptoms

DETAILED DESCRIPTION:
Background: Prevalence of endometriosis is approximately 10% of women of childbearing age. Pain, considered in its multiple versions (dysmenorrhea, dyspareunia, dyschezia, dysuria and, in general, chronic pelvic pain) is the most common and disabilitating symptom in affected women. Usual care, consisting on palliative pharmacological treatment in combination with surgery, is clearly insufficient and physical therapies need to be explored in order to reduce pain and to improve quality of life in affected women.

Objective: The overall objective of 'Physio-EndEA' study will be to explore potential short and mid-term benefits of a rehabilitation program on the quality of life of symptomatic women.

Methods: A total of 26 symptomatic endometriosis women will be recruited. Inclusion criteria includes: aged 18-50, clinical diagnosis of endometriosis and interested in improving lifestyle while exclusion criteria includes: diagnosed chronic disease or orthopaedic issues that would interfere with ability to participate in a physical activity program. Women will be randomized to either intervention (n=13) or usual care group (n=13). Intervention group will receive twice weekly session for 9 weeks and control group will receive recommendations about healthy lifestyle and usual care.

Discussion: This study attempts to improve the quality of life of symptomatic endometriosis women by reducing musculoskeletal and occupational impairments. Findings will offer a new therapeutic approach for a better pain control.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal status
* Clinical diagnosis of endometriosis by laparoscopy, magnetic resonance imaging or ultrasound imaging
* History of clinical symptoms
* To be able to walk without assistance
* To be able to read and write enough
* To be capable and willing to provide consent
* Interested in improving lifestyle

Exclusion Criteria:

* Acute or terminal illness
* Presence of any chronic disease or orthopedic issues that would interfere with ability to participate in a physical activity program
* Unwillingness to complete the study requirements
* Be registered in other exercise program

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life assessed by EHP-30 | Baseline, inmediately after intervention and 1-year post-intervention
  It will be assessed using the Endometriosis Health Profile-30 (EHP-30). It is a self-administered disease-specific instrument to measure QoL in women with endometriosis. The 30-item EHP, referred to the last 4 weeks, is comprised of five domains: pain, control and powerlessness, emotional well-being, social support, and self-image. Items within each subscale, answered on a 5-point Likert-type scale, are summed and then transformed to a percentage scale ranging from 0 (best health status) to 100 (worse health status) by dividing the raw score of all items by the maximum possible raw score, multiplied by 100

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | Baseline, inmediately after intervention and 1-year post-intervention
  Algometry will be used to measure PPT levels in abdomen, pelvis and lower back regions through an electronic algometer. For this purpose, an approximate rate of 30 kilopascal/s will be applied with a 1cm2 probe. Seven points from the abdominal and pelvic area, and two additional points from the lower back region will be tested. Prior PPT assessment, assessor will ask for participants to press the switch when they first feel a change from pressure to pain. The mean of three tests, spaced by 30 s, will be used for the analysis.
Pain intensity | Baseline, inmediately after intervention and 1-year post-intervention
  Visual Analogue Scale will be used to identify self-reported levels of chronic pelvic pain, dysmenorrhea, dyspareunia, dyschezia and dysuria.. Scores range from 0 to 10. Higher scores represent increased pain intensity
Catastrophizing thoughts | Baseline, inmediately after intervention and 1-year post-intervention
  The Pain Catastrophizing Scale (PCS) will be also used to assess catastrophic thinking related to pain. Scores of this 13-item scale range from 0 to 52. Higher scores represent higher catastrophic thoughts.
Muscle thickness | Baseline, inmediately after intervention and 1-year post-intervention
  Images of the abdominal wall, lumbar multifidus and quadriceps will be obtained using an ultrasound device with a 12 megahertz linear probe and a depth of 5 cm. The thicknesses of the external and internal oblique, the transversus abdominal muscles and the lumbar multifidus, as well as the width of the lumbar multifidus will be assessed. Three measurements of both right and left muscles diameters will be recorded with a 2-minute interval between trials.
  Lumbar multifidus assessment will be performed at, the fifth lumbar vertebra, marking its spinal process.
Muscle trunk flexor and extensor endurance | Baseline, inmediately after intervention and 1-year post-intervention
  Muscle trunk flexor endurance test will be used to assess the endurance strength of abdominal muscles by isometric endurance of trunk flexors. Time (in seconds) is measured, and higher scores represent better performance.
  Muscle trunk extensor endurance test will be used to assess the endurance strength of back extensor muscles by isometric endurance of trunk extensors.Time (in seconds) is measured, and higher scores represent better performance.
Flexibility of the lumbar spine | Baseline, inmediately after intervention and 1-year post-intervention
  Original Schöber test will be used to assess lumbar spine flexibility. The assessor will determine the location of the lumbosacral junction and marks it with a horizontal line. A second mark will be drown 10cm above the first line. The difference between the measurements in erect and flexion positions will be recorded. Higher differences represent better flexibility.
Body Balance | Baseline, inmediately after intervention and 1-year post-intervention
  Total body balance will be assessed with the Flamingo test. In standing position without shoes, participants will be asked to stay on one leg. Assessor will record the number of trials needed to complete 30 seconds of this static position. The average of both legs will be used. Lower scores represent better performance
Functional capacity | Baseline, inmediately after intervention and 1-year post-intervention
  It will be assessed with theThe 6-min walk test (6MWT) to determine the maximum distance that each patient is able to walk within 6 min (in metres). Patients are instructed to walk as far as they can in 6 min, without stopping and without running, but increasing and decreasing the speed voluntarily. Higher scores represent better performance
Chronic fatigue | Baseline, inmediately after intervention and 1-year post-intervention
  Muscular fatigue will be assessed with the Piper Fatigue Scale-Revised (PFS-R), originally developed to assess cancer-related fatigue, but also used to assess fatigue in other musculoskeletal disorders such as heart failure. It contains 22 items scoring from 0 to 10. Total score is average score of these 22 items (0-10). Lower scores reflect better performance. PFS-R has high reliability (Cronbach's α=0.96).
Body mass index | Baseline
  Height (in centimeters) and weight (in kilograms) will be assessed and then combined to report body mass index (BMI) in kg/m^2.
Skeletal muscle mass | Baseline
  Skeletal muscle mass (in kilograms) will be recorded with an impedance meter
Body fat | Baseline
  Body fat (in percentage) will be recorded with an impedance meter
Sexual function | Baseline, inmediately after intervention and 1-year post-intervention
  It will be assessed with the Female Sexual Function Index questionnaire (FSFI) (19 item) divided in 6 domains:desire, arousal, lubrication, orgasm, satisfaction and pain.
  Items are answered on a 6-point Likert-type scale (with the exception of items 1 and 2, answered on a 5-point Likert-type scale). Scores of individual items from each domain are summed and multiplied by the domain factor. The global score is obtained by the sum of all domain scores, ranging from 2 to 36. Higher values correspond to better sexual function
Gastrointestinal function | Baseline, inmediately after intervention and 1-year post-intervention
  It will be assessed with the Gastrointestinal Quality of Life Index (GLQI) (36 items) grouped in 5 domains: digestive symptoms, physical status, emotions, social dysfunction and effects of medical treatment. Each item is scored from 0 (worst appreciation) to 4 (best appreciation). Scores of items are summed to obtain the global score, which ranges from 0 (worst) to 144 (best quality of life).
Sleep quality | Baseline, inmediately after intervention and 1-year post-intervention
  It will be assessed with the Pittsburgh Sleep Quality Index (PSQI) (19 items), grouped in seven "components": subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component ranges from 0 (lowest dysfunction) to 3 (greatest dysfunction), and the PSQI global score is obtained by the sum of component's scores, and thus, ranges from 0 to 21, with higher scores indicating poor sleep quality.
Self-perceived physical fitness | Baseline
  Regular physical activity will be estimated through the Minnesota Leisure Time Physical Activity Questionnaire (MLTPAQ), that has shown a moderate reliability to indirectly estimate physical activity (Spearman rank correlation coefficient > 0.69). During an interview, the assessor will ask each women the number of days per week and the amount of time (in minutes) per day that they spent doing each of the 63 activities listed in the questionnaire. Finally, an activity metabolic index is calculated by multiplying the number of days per week, the amount of time per day and the standard intensity codes assigned to each activity. This score approximates Kcal/day of energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Artacho-Cordón, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Francisco Artacho Cordón, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salinas-Asensio MDM, Alvarez-Salvago F, Mundo-Lopez A, Ocon-Hernandez O, Lozano-Lozano M, Lopez-Garzon M, Postigo-Martin P, Arroyo-Morales M, Rodriguez-Ruiz A, Fernandez-Lao C, Artacho-Cordon F. Changes in fatigue, health-related fitness, sleep quality, mental health, gastrointestinal complaints and sexual function after a multimodal supervised therapeutic exercise program in women with endometriosis unresponsive to conventional therapy: a secondary analysis of a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2025 Aug;312:114083. doi: 10.1016/j.ejogrb.2025.114083. Epub 2025 May 24. PMID 40440865
- [Derived] Artacho-Cordon F, Salinas-Asensio MDM, Galiano-Castillo N, Ocon-Hernandez O, Peinado FM, Mundo-Lopez A, Lozano-Lozano M, Alvarez-Salvago F, Arroyo-Morales M, Fernandez-Lao C, Cantarero-Villanueva I. Effect of a Multimodal Supervised Therapeutic Exercise Program on Quality of Life, Pain, and Lumbopelvic Impairments in Women With Endometriosis Unresponsive to Conventional Therapy: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Nov;104(11):1785-1795. doi: 10.1016/j.apmr.2023.06.020. Epub 2023 Jul 17. PMID 37467936